CLINICAL TRIAL: NCT03350984
Title: Insulin Scheme for Glycemic Control in Non-critical Hospitalized Patients With Type 2 Diabetes in the Context of a Health System in Mexico.
Brief Title: Insulin Schemes for Type 2 Diabetes Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Jose Antonio de Jesus Alvarez Canales, PhD, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSGTO00136
Record Dates: First submitted 2017-11-06; First posted 2017-11-22 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin, Isophane; Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NPH insulin group (Experimental): Patients receiving NPH twice daily, 2/3 in the morning and 1/3 in the night. A correctional dose of lispro insulin will be given for any blood glucose >180 mg/dL. If subjects were not eating, they shouldn't receive dose of NPH insulin. Intervention Drug: NPH insulin
  Interventions: Drug: NPH insulin
- Glargine and Lispro insulin group (Active Comparator): Half of the total of Glargine and Lispro insulin dose will be given as glargine once daily, either in the morning or in the evening, depending on when the patient was enrolled. The other half of the total daily insulin dose will be given as Lispro; doses were divided equally for breakfast, lunch, and dinner. An additional correctional dose of Lispro will be given for any blood glucose >180 mg/dL. If subjects were not eating, they received glargine once daily and they shouldn't receive doses of lispro.
  Intervention drug: Glargine and Lispro
  Interventions: Drug: Glargine and Lispro insulin

INTERVENTIONS:
Drug: NPH insulin — NPH insulin twice daily, 2/3 in the morning and 1/3 in the night. A correctional dose of lispro insulin will be given for any blood glucose >180 mg/dL.
  Other Names: NPH
  Arms: NPH insulin group
Drug: Glargine and Lispro insulin — Half of the total Glargine and Lispro insulin dose will be given as glargine once daily, either in the morning or in the evening, depending on when the patient was enrolled. The other half of the total daily insulin dose was given as Lispro; doses were divided equally between breakfast, lunch, and dinner.
  Other Names: Glargine and Lispro
  Arms: Glargine and Lispro insulin group

SUMMARY:
The aim of the study is to determine differences in glycemic control between a basal-bolus scheme insulin and NPH scheme insulin in a population of hospitalized patients with type 2 diabetes in a Noncritical Care Facility in Mexico. Patients with a recent diagnosis of type 2 and patients on treatment with oral hypoglycaemic agents and insulin or only insulin were included.

The primary outcome of the study is to determine difference in efficacy and security between a basal-bolus scheme insulin and NPH scheme insulin in patients with type 2 diabetes hospitalized in non-critical areas in a hospital in Mexico

DETAILED DESCRIPTION:
On the first 4 to 6 h, the use of NPH insulin present a pronounced action peak on the postprandial glucose metabolism, and the rest of its basal action last 12 to 18 h, its cover the postprandial requirements of the first two meals of the day (breakfast and lunch) administering 2/3 of the total dose, and the requirements for the dinner with 1/3 of the total dose at the night. This is considered a good scheme for handling hyperglycemia, and its possible to have less hypoglycemia episodes, which are possible if an ultra-rapid-acting insulin is added and adequate intake is not performed due to multiple factors related to hospitalization.

Today it is uncertain whether there is any clear benefit of using Glargine plus Lantus insulin over NPH insulin in hospitalized patients with type 2 diabetes. Currently, both Glargine and NPH based regimen is practiced in inpatient hospital facilities. Current practice of inpatient insulin regimen is based on the physicians familiarity with a particular insulin type and personal preference rather than evidenced based knowledge. Glargine plus ultrafast insulin are two types of insulin that are more expensive compared to NPH with incidental benefits in hospitalized patients. There are reports in the literature about the incidence of hypoglycemia with this scheme. The current research proposal is to compare these two schemes in the treatment of hospitalized patients with diabetes in a hospital of the second level of care in Mexico.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 100 years old.
* History of type 2 diabetes mellitus (DM2) or that upon admission is diagnosed by values of glycated haemoglobin (HbA1) > 6.5%
* Fasting central glucose before randomization between 140mg/dl and 400mg/dl
* Non-critical patients hospitalized in the service of Internal Medicine (MI), General Surgery (CG) and Traumatology (TyO).
* Patients receiving a diabetic diet orally
* Treated with diet alone, o any combination of oral anti-diabetic agents or insulin treatment with any dosage before admission.

Exclusion Criteria:

* Parenteral nutrition
* Hyperglycemia without a known history of diabetes
* Impaired renal function (glomerular filtration rate less than 30)
* Diabetic ketoacidosis and hyperosmolar state
* Type 1 Diabetes mellitus
* Pregnancy
* Patients on treatment with more than 10mg prednisone or steroid boluses.
* Known hypopituitarism or adrenal insufficiency
* Hyperglycaemia due to stress (negative antecedent of DM2, hyperglycemia and HbA1 <6.5)
* Severe liver disease (Child-Pugh C score)
* Acute pancreatitis
* Patients with sepsis or multiple organ failure
* Candidates for intensive care unit

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Alvarez, PhD, Principal Investigator — Universidad de Guanajuato
Locations (1):
- Hospital General de León, León, Guanajuato, Mexico

REFERENCES:
- [Background] Umpierrez GE, Smiley D, Jacobs S, Peng L, Temponi A, Mulligan P, Umpierrez D, Newton C, Olson D, Rizzo M. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes undergoing general surgery (RABBIT 2 surgery). Diabetes Care. 2011 Feb;34(2):256-61. doi: 10.2337/dc10-1407. Epub 2011 Jan 12. PMID 21228246
- [Background] Umpierrez GE, Smiley D, Hermayer K, Khan A, Olson DE, Newton C, Jacobs S, Rizzo M, Peng L, Reyes D, Pinzon I, Fereira ME, Hunt V, Gore A, Toyoshima MT, Fonseca VA. Randomized study comparing a Basal-bolus with a basal plus correction insulin regimen for the hospital management of medical and surgical patients with type 2 diabetes: basal plus trial. Diabetes Care. 2013 Aug;36(8):2169-74. doi: 10.2337/dc12-1988. Epub 2013 Feb 22. PMID 23435159
- [Background] Christensen MB, Gotfredsen A, Norgaard K. Efficacy of basal-bolus insulin regimens in the inpatient management of non-critically ill patients with type 2 diabetes: A systematic review and meta-analysis. Diabetes Metab Res Rev. 2017 Jul;33(5). doi: 10.1002/dmrr.2885. Epub 2017 Feb 23. PMID 28067472

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 111 hospitalized DM2 patients not critical to the study were evaluated. Of these, 35 did not meet the inclusion criteria and the 75 included participants were randomized into two groups. The recruitment of patients began on November 2, 2017 and ended on June 1, 2018.
Pre-assignment Details: Within the basal-bolus group, 1 patient was eliminated before initiating the insulin regimen, presenting acute abdomen and requiring intensive therapy. Therefore, 36 patients will start treatment in the basal-bolus group and 39 patients in the NPH group.
Groups:
- Glargine and Lispro Insulin Group: Half of the total of Glargine and Lispro insulin dose will be given as glargine once daily, either in the morning or in the evening, depending on when the patient was enrolled. The other half of the total daily insulin dose will be given as Lispro; doses were divided equally for breakfast, lunch, and dinner. An additional correctional dose of Lispro will be given for any blood glucose >180 mg/dL. If subjects were not eating, they received glargine once daily and they shouldn't receive doses of lispro.
  Intervention drug: Glargine and Lispro
  Glargine and Lispro insulin: Half of the total Glargine and Lispro insulin dose will be given as glargine once daily, either in the morning or in the evening, depending on when the patient was enrolled. The other half of the total daily insulin dose was given as Lispro; doses were divided equally between breakfast, lunch, and dinner.
Period: Overall Study
Arm/Group | NPH Insulin Group | Glargine and Lispro Insulin Group
Started | 39 | 36
Completed | 31 | 28
Not Completed | 8 | 8
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 5 | 6
Not completed — Protocol Violation | 1 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NPH Insulin Group | Glargine and Lispro Insulin Group | Total
Number analyzed (Participants) | 39 | 36 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 27 | 52
  >=65 years | 14 | 9 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13.1) | 56.4 (12.9) | 57.8 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 19 | 15 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 36 | 75
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 39 | 36 | 75
Central glucose [Mean (Standard Deviation); unit: mg / dl] — Measurement of central glucose levels on admission (mg/dl).
  mg / dl | 237.3 (73.1) | 223.1 (67) | 230.5 (70.2)

OUTCOME MEASURES:

1. Primary Outcome: Differences in the Mean Daily Blood Glucose Between a Basal-bolus Scheme and NPH Schemes of Insulin.
Description: To determine the differences in the mean daily blood glucose measured in mg/dl, between a basal-bolus scheme and NPH schemes of insulin measured by the mean daily blood glucose.
Time Frame: Fasting blood glucose was taken every day, before breakfast, up to 4 weeks; postprandial glucose was taken every day, 2 hours after breakfast, 2 hours after lunch, and 2 hours after dinner, up to 4 weeks; glucose early morning was taken 3 am, up to 4 week
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | NPH Insulin Group | Glargine and Lispro Insulin Group
Number analyzed (Participants) | 39 | 36
mg/dl
  Fasting blood glucose | 129.6 (23.6) | 135 (22.6)
  Postprandial glucose | 155.4 (29) | 156.2 (27.2)
  Glucose in the early morning | 127.4 (26.6) | 136.2 (21.2)

2. Secondary Outcome: the Number of Participants With Mild and Severe Hypoglycemic Events
Description: To measure the number of participants with mild and severe hypoglycemic events
Time Frame: Duration of hospital stay, up to 4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | NPH Insulin Group | Glargine and Lispro Insulin Group
Number analyzed (Participants) | 39 | 36
Participants | 15 | 15

3. Secondary Outcome: Number of Participants With Sustained Glycemic Control During Hospital Stay
Description: Sustained glycemic control were the number of participants who not had: discharged before sustained control, critical status suspension, death before control, bad attachment to the protocol, interruption due to more than 2 hypoglycemic events during their hospital stay.
Time Frame: blood glucose was taken every day, up to 4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | NPH Insulin Group | Glargine and Lispro Insulin Group
Number analyzed (Participants) | 39 | 36
Participants | 30 | 20

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | NPH Insulin Group | Glargine and Lispro Insulin Group
All-Cause Mortality (participants affected / at risk) | 1/39 | 1/36
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/36
Other Adverse Events (participants affected / at risk) | 15/39 | 11/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPH Insulin Group (N=39) | Glargine and Lispro Insulin Group (N=36)
Soft tissue infection (Infections and infestations) | 14 (14) | 9 (9)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Although the patients had an oral diet, the prolonged stay due to complications not associated with DM2 reduced their caloric intake.

The physiological scheme is more demanding, making it difficult to stick to the ideal conditions of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT03350984/Prot_SAP_ICF_000.pdf